CLINICAL TRIAL: NCT05202080
Title: Effect of a Pre-operative Internet-based Educational Video, Providing Both Opioid Counselling and Pain Coping Skills, on Post-operative Opioid Consumption
Brief Title: Effect of a Pre-operative Internet-based Educational Video on Post Operative Opioid Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ahtsham Niazi, Associate Professor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5218
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Patient Empowerment
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Counseling and PCS Video Group (Experimental): This arm of the study will receive the opioid counseling and pain coping skills video 2 weeks prior to their surgery in addition to the conventional information provided to all patients undergoing total joint arthroplasty.
  Interventions: Other: Opioid Counseling and Pain Coping Skills Video
- Standard of Care Group (No Intervention): This arm of the study will the conventional information provided to all patients undergoing total joint arthroplasty.

INTERVENTIONS:
Other: Opioid Counseling and Pain Coping Skills Video — The intervention will be in the form of a video of a PowerPoint presentation with instructions and exercises designed to coach patients about catastrophizing, coping skills, mindfulness and behavioral modification techniques, in addition to providing education regarding postoperative analgesia and opioid use.
  Arms: Opioid Counseling and PCS Video Group

SUMMARY:
One of the most challenging issues in modern medicine is the current opioid epidemic. Given the association between opioid use after surgery and the development of opioid addiction, an essential goal of the medical community should be to develop strategies aimed at instructing the safe use of opioids. In addition, instructions on how to use non-opioid painkillers and exercises and techniques to better cope with pain can be used to reduce the patients opioid requirements after surgery. This study aims to evaluate the effect of providing an online educational video presentation to patients prior to surgery. This will be a 30 minute video which will provide the study participants with instructions on how best to use their opioid and non-opioid medication for pain and also teach the study participants exercises and techniques to better cope with their pain. This intervention will be used with a view to reduce the amount of opioids used by patients following hip or knee replacement surgery. Participants will be followed during their immediate phase after surgery to determine how much pain killers the participants have used and at six weeks the participants will be asked to return their unused opioids to see how much the participants have used in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adults (> 18 years of age) undergoing knee or hip arthroplasty.
* Patients will be ASA 1-3 undergoing elective surgery.
* English speaking patients with internet and computer access at home will be included.
* Patients with pre-existing psychological conditions who receive either pharmaceutical or talk-based therapy will be included.
* Patients must meet a minimum cognitive capacity to understand the instructions for the Opioid Counseling and Pain Coping Skills presentation. This will be assessed by the administration of the Montreal Cognitive Assessment during screening (MoCA), whereby a minimum score of 18 will be required to meet inclusion into the study.

Exclusion Criteria:

* Significant cognitive impairment.
* Chronic pain, long-term opioid therapy
* Renal replacement therapy
* Standing opioid requirements
* Neuropathic pain
* Fractures requiring emergency surgery
* End stage cardiac or respiratory disease
* Severe hepatic dysfunction,
* Patients with severe psychiatric disorders
* Vision loss
* Allergy to local anesthesia.
* Patients who refuse to consent to neuraxial anesthesia and/or peripheral nerve blocks will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Post operative opioid consumption | 2 weeks postoperatively
  opioid tablets used in the 2 weeks post operatively

SECONDARY OUTCOMES:
Postoperative Pain | 72 hours post operatively
  Using the Verbal Analog Scale (VAS) for Pain Assessment from 0 to 10 with 0 being no pain and 10 being extreme pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No